CLINICAL TRIAL: NCT00499265
Title: A Randomized, Open Label, Phase II Proof of Concept Study of WX-671 in Combination With Gemcitabine vs.Gemcitabine Alone in Patients With Locally Advanced, Non Resectable Pancreatic Cancer in Order to Evaluate the Anti-Tumor Activity of the Combination Therapy
Brief Title: Gemcitabine With or Without WX-671 in Treating Patients With Locally Advanced Pancreatic Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000553460; WILEX-WX-60-004
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; upamostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gemcitabine (Active Comparator)
  Interventions: Drug: gemcitabine hydrochloride
- Gemcitabine plus 200 mg WX-671 (Experimental)
  Interventions: Drug: Serine Proteinase Inhibitor WX-671
- Gemcitabine plus 400 mg WX-671 (Experimental)
  Interventions: Drug: Serine Proteinase Inhibitor WX-671

INTERVENTIONS:
Drug: gemcitabine hydrochloride — 1000 mg/m2 as 30 min i.v. infusion once weekly for 7/8 weeks and then every 3/4 weeks
  Other Names: GEMZAR
  Arms: Gemcitabine
Drug: Serine Proteinase Inhibitor WX-671 — oral, daily
  Other Names: MESUPRON
  Arms: Gemcitabine plus 200 mg WX-671
Drug: Serine Proteinase Inhibitor WX-671 — oral, daily
  Other Names: MESUPRON
  Arms: Gemcitabine plus 400 mg WX-671

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. WX-671 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving gemcitabine together with WX-671 may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying how well gemcitabine works when given together with WX-671 or when given alone in treating patients with locally advanced pancreatic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the antitumor activity of two different doses of anti-uPA serine protease inhibitor WX-671 when given in combination with gemcitabine hydrochloride in patients with locally advanced unresectable pancreatic cancer.
* Compare the efficacy, in terms of response rate, progression-free survival, time to first metastasis, overall survival, and tumor and uPA system-related markers, of these regimens in these patients.
* Compare the safety, in terms of vital signs, ECG, biochemistry, hematology (including coagulation), and adverse events, of these regimens.

OUTLINE: This is an open-label, randomized, multicenter study. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive of oral anti-uPA serine protease inhibitor WX-671 once daily in weeks 1-8 (weeks 1-4 of each subsequent course) and gemcitabine hydrochloride IV over 30 minutes once weekly in weeks 1-7 (weeks 1-3 of each subsequent course) of course 1. All subsequent courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral anti-uPA serine protease inhibitor WX-671 (at a lower dose than in arm I) once daily in weeks 1-8 (weeks 1-4 of each subsequent course) and gemcitabine hydrochloride IV over 30 minutes once weekly in weeks 1-7 (weeks 1-3 of each subsequent course) of course 1. All subsequent courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
* Arm III: Patients receive gemcitabine hydrochloride IV over 30 minutes once weekly in weeks 1-7 (weeks 1-3 of each subsequent course) of course 1. All subsequent courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Inclusion criteria:

  * Locally advanced, unresectable, non-metastatic, histologically proven pancreatic adenocarcinoma (lymph nodes will not be considered metastases)
* Exclusion criteria:

  * Any distant metastases

PATIENT CHARACTERISTICS:

* Inclusion criteria:

  * ECOG performance status ≤ 1
  * Life expectancy > 12 weeks
  * Normal 12-lead ECG or only clinically insignificant abnormalities in the judgment of the investigator
  * Female patients of child-bearing potential will be required to use an effective method of birth control for the duration of the study to prevent pregnancy
  * ANC ≥ 1,500/mm³
  * Platelet count ≥ 100,000/mm³
  * Hemoglobin ≥ 9 g/dL
  * Total bilirubin ≤ 1.5 times ULN
  * AST and ALT ≤ 2.5 times ULN
  * Alkaline phosphatase ≤ 2.5 times ULN
  * Creatinine ≤ 2 times ULN or creatinine clearance > 45 mL/min
* Exclusion criteria:

  * History of or current primary blood coagulation or bleeding disorders such as hemophilia
  * Any unrelated illness, e.g., active infection, inflammation, medical condition or laboratory abnormalities, which in the judgment of the investigator might significantly affect the patient's study participation
  * Any surgical or medical condition that might significantly alter the absorption, distribution, metabolism or excretion of any drug
  * Significant cardiac insufficiency (NYHA classification III or IV), presence of unstable angina or myocardial infarction within the previous 6 months, use of ongoing maintenance therapy for life threatening arrhythmia or known pulmonary hypertension
  * Any secondary malignancies within the last 5 years except for surgically cured non-melanoma skin cancer or cervical carcinoma in situ
  * Pregnancy (positive serum pregnancy test) or lactation
  * Known hepatitis B/C or HIV infection
  * Known hypersensitivity to any of the components in the anti-uPA serine protease inhibitor WX-671 capsules or gemcitabine hydrochloride infusion or other medical reasons for not being able to receive adequate pre-medication (for example, antihistamine or anti-inflammatory agents)

PRIOR CONCURRENT THERAPY:

* Permitted:

  * Growth factors for treatment (not prophylaxis, i.e., epoetin alfa), analgesics, blood transfusions, antibiotics, bisphosphonates, other hormonal therapy for contraceptive practice, replacement therapy such as thyroid replacement or adrenal insufficiency as appropriate and medications for acute or chronic conditions not listed under the exclusion criteria
  * Embolization (i.e. for hematuria)
  * Subjects can receive blood transfusions as medically appropriate during the study

    * Subjects who require a blood transfusion during screening must have stable hemoglobin (≥9.0 g/dL [5.6 mmol/L]) without the need for further transfusions within 2 weeks before the first dose of anti-uPA serine protease inhibitor WX-671 to remain eligible
  * Prophylactic use of growth factors to support neutrophils
* Prohibited:

  * Anticoagulant or thrombolytic therapy within four weeks prior to start of treatment (except low dose anticoagulant therapy with unfractionated heparin ≤ 15000 IU/d, low molecular weight heparin ≤ 5000 IE anti-Xa activity or acetyl salicylic acid ≤ 100 mg/d at the discretion of the investigator)
  * Anticancer therapies such as biologic therapy and chemotherapy (other than study drugs)
  * Radiation therapy (during the treatment phase of the protocol; increased bone pain not controlled by medication and requiring palliative therapy will be considered disease progression)
  * Laser treatment
  * Any other investigational agent
  * Thalidomide
  * Immunosuppressive therapies (inhaled or replacement dose corticosteroids are permitted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2007-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Efficacy, in terms of response rate, progression-free survival, time to first metastasis, overall survival, and tumor and uPA system-related markers | 3 years
Safety, in terms of vital signs, ECG, biochemistry, hematology (including coagulation), and adverse events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Carola Mala, PhD, Study Chair — Heidelberg Pharma AG
Locations (39):
- Germany (9):
  - Charite University Hospital - Campus Virchow Klinikum, Berlin
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Otto-Meyerhof-Zentrum Tagesklinik, Heidelberg
  - Universitaetsklinkum Magdeburg der Otto-von-Guericke-Universitaet Magdeburg, Magdeburg
  - Johannes Gutenberg University, Mainz
  - III Medizinische Klinik Mannheim, Mannheim
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Hospital Muenchen Bogenhausen, Munich
- Hungary (5):
  - Szent Laszlo Korhaz, Budapest
  - Debreceni Egyetem Onkologiai Tanzek, Debrecen
  - Petz Aladar County Hospital, Gydr
  - University of Pecs Faculty of Medicine, Pécs
  - Szeged University, Szeged
- Italy (5):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Presidio Ospedaliero di Livorno, Livorno
  - Azienda Ospedaliera di Rilievo Nazionale A.Cardarelli, Naples
  - Istituto Tumori/Fondazione Pascale, Naples
  - Ospedale San Filippo Neri, Rome
- Russia (7):
  - Altai Oncology Center, Barnaul
  - Moscow Oncology Hospital, Moscow
  - Russian Academy of Medical Sciences Cancer Research Center, Moscow
  - Central Clinical Hospital of the President of the Russian Federation, Moscow
  - Rostov Research Institute of Oncology - Omsk, Omsk
  - Pavlov State Medical University, Saint Petersburg
  - Saint Petersburg State Medical University, Saint Petersburg
- Spain (5):
  - Hospital de la Santa Cruz i Sant Pau, Barcelona
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Universitario de Elche, Elche
  - Hospital Virgen de las Nieves, Granada
  - Centro Oncologico M.D. Anderson International Espana, Madrid
- Ukraine (8):
  - Cherkassy Regional Oncology Center, Cherkassy
  - Bukovinian State Medical University, Chernivtsy
  - Dnipropetrovsk State Medical Academy, Dnipropetrovsk
  - Donetsk Regional Antitumor Center, Donetsk
  - Ivano-Frankovsk Regional Oncology Center, Ivano-Frankivsk
  - Grigoriev Institute for Radiology Academy of Medical Science of Ukraine, Kharkiv
  - Institute of Oncology, Kiev
  - Ukrainian Medical Stomatological Academy, Poltava